CLINICAL TRIAL: NCT06694506
Title: BELux Children OutcoME During A(@)Dulthood With Growth Hormone Deficiency
Brief Title: BELux Children OutcoME During A(@)Dulthood With GHD
Acronym: BELCOME@GHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CUSL
Record Dates: First submitted 2024-07-25; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Growth Hormone Deficiency; Adult Growth Hormone Deficiency
Keywords: Growth Hormone; Adult
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Intervention Model Description: We aim to include both male and female adult patients with a diagnosis of childhood onset-GHD, registered in BELGROW, that stopped the GH therapy for growth after 2011 and have a persistent GHD in adolescence/transition period. After completing a questionnaire, each participant will be assigned an analysis group:
  * Group 1: Patients with regular follow-up for their GHD (treated with rhGH or not) in a adult endocrinology department including a clinical examination and endocrine blood work-up at least once a year
  * Group 2: Patients who are lost to follow-up or not regularly followed for their GHD (or only followed by their GP with no endocrine assessment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with regular follow-up for their GHD (treated with rhGH or not) (No Intervention): Patients with regular follow-up for their GHD (treated with rhGH or not) in a adult endocrinology department including a clinical examination and endocrine blood work-up at least once a year
- Patients who are lost to follow-up or not regularly followed for their GHD (Active Comparator): Patients who are lost to follow-up or not regularly followed for their GHD (or only followed by their GP with no endocrine assessment)
  Interventions: Other: Biological Sample

INTERVENTIONS:
Other: Biological Sample — Clinical examination and blood test. The clinical examination and blood test are considered standard-of-care as they could be performed annually or bi-annually as part of an adult GHD follow-up. Subsequently, the data will be collected directly from the patient's chosen physician.
  Arms: Patients who are lost to follow-up or not regularly followed for their GHD

SUMMARY:
Our objective is to evaluate the outcome in adulthood of Belgian and Luxembourgish patients treated with rhGH during childhood for CO-GHD. The primary goal is to determine the proportion of adult CO-GHD patients who continue to receive regular medical follow-up and those still undergoing rhGH therapy using a questionnaire. Secondary objectives include assessing the regularity of follow-up and compliance with treatment in adulthood, evaluating possible comorbidities, health issues, lifestyle, living environment, and quality of life. Additionally, we aim to assess the metabolic profile in adulthood, particularly focusing on BMI, glycemic, and lipid data, for patients who consent to share their current clinical and biological data. Data will be described according to treatment adherence and CO-GHD etiology/phenotypes (e.g., idiopathic vs. organic GHD, isolated vs. combined GHD, partial vs. severe GHD).

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Diagnosed with child-hood onset growth hormone deficiency (CO-GHD) (no exclusion criteria: isolated or multiple GHD, idiopathic or organic, severe or partial)
* Registered in the BELGROW registry (informed consent at the time of inclusion in registry)
* Stopped treatment with rhGH for growth after 2011
* Persistent GHD at the end of growth

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Determine the proportion of adult CO-GHD patients who continue to receive regular. medical follow-up | Baseline
  Using our questionnaire, the primary objective is to determine the proportion of adult CO-GHD patients who continue to receive regular medical follow-up (and where/by who) and the proportion of patients still undergoing rhGH therapy.

SECONDARY OUTCOMES:
Assessment of the regularity of follow-up and compliance with a questionnaire. | Baseline
  Assessment of the regularity of follow-up and compliance to treatment in adulthood (in patients that are still followed and/or treated with rhGH therapy), with the help of a questionnaire created by the research team.
Assessment of the possible comorbidities and health issues with a questionnaire. | Baseline
  Assessment of the possible comorbidities and health issues, lifestyle, living environment and quality of live (all patients) in adulthood. with the help of a questionnaire created by the research team.
Assessment of the metabolic profile in adulthood. | 1 year per patient
  Assessment of the metabolic profile in adulthood - particularly in relation to BMI, glycemic and lipid data. (fasting glycemia, fasting insulin, hemoglobin A1c, transaminase levels, lipid profile (total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides), insulin-like growth factor 1 (IGF-1) levels, and other hormone levels (thyroid-stimulating hormone (TSH), thyroxine (T4), prolactin (PRL), luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol/testosterone, cortisol).). Each of these data will be compared with the clinical data in the same way.
Describe those data according to treatment adherence. | Baseline
  Describe those data according to treatment adherence and CO- GHD etiology/phenotypes (e.g. idiopathic vs organic GHD, isolated vs combined GHD, partial vs severe GHD) The questionnaire will provide us with information on patients' adherence to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Woluwe-saint-lambert, Belgium

IPD SHARING:
Plan to Share IPD: No